CLINICAL TRIAL: NCT05860491
Title: The Role of Dietary Fiber on Hyperkalemia in Hemodialysis Patients
Brief Title: Dietary Fiber and Hyperkalemia in Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Yang Li, Attending physician, Qianfoshan Hospital
Other Study IDs: DF-hyperkalemia
Record Dates: First submitted 2023-05-08; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Hyperkalemia; Hemolysis
MeSH Terms: conditions — Hyperkalemia; Hemolysis | interventions — Dietary Fiber

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with pre-dialysis hyperkalemia: To investigate the dietary fiber intake of hemodialysis patients with pre-dialysis hyperkalemia. Use a retrospective analysis method. Analyze the relationship between dietary fiber intake and hyperkalemia.
  Interventions: Other: dietary fiber
- patients without pre-dialysis hyperkalemia: To investigate the dietary fiber intake of hemodialysis patients without pre-dialysis hyperkalemia. Use a retrospective analysis method. Analyze the relationship between dietary fiber intake and hyperkalemia.
  Interventions: Other: dietary fiber

INTERVENTIONS:
Other: dietary fiber — Retrospective analysis of the relationship between patient dietary fiber intake and hyperkalemia

SUMMARY:
To analyze the dietary nutrition and dietary fiber (DF) intake of maintenance hemodialysis (MHD) patients, and explore the effect of dietary nutrition and DF intake balance on the nutritional status and pre-dialysis hyperkalemia of MHD patients.

DETAILED DESCRIPTION:
A total of 100 MHD patients were retrospectively enrolled, including 67 males and 33 females. The daily diet was recorded by 3-day dietary recording method. The daily average dietary nutritional intake and DF intake of MHD patients were calculated by professional software. Dietary guidance and analysis were conducted according to the Expert Consensus on Nutrition in Chronic Kidney Disease (2005) and the Dietary Guidelines for Chinese Residents (2016). Of the 100 patients, 37 had hyperkalemia (serum potassium > 5.5 mmol/L) before dialysis.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old; undergoing hemodialysis at least 3months; with a certain level of education; with complete behavioral ability

Exclusion Criteria:

* In the acute phase of acute cardiovascular disease, acute cerebrovascular disease, and acute digestive system disease；Anorexia, long-term malnutrition, or dietary disorders；poor compliance；

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing hemodialysis
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Dietary fiber intake | 3 day
  Dietary fiber intake

CONTACTS AND LOCATIONS:
Overall Officials: Yang Li, Master, Principal Investigator — Qianfoshan Hospital
Locations (1):
- Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided
undecided